CLINICAL TRIAL: NCT03826511
Title: The Effects of Tiszasüly and Kolop Mud-pack Therapy in Knee Osteoarthritis: Randomized Non-inferiority Controlled Pilot Study
Brief Title: The Effects of Tiszasüly and Kolop Mud-pack Therapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Principal Investigator, Márta Király, chief physician, Petz Aladar County Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PetzCTH
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
Keywords: mud-pack therapy; osteoarthritis of the knee; hot-pack therapy; non-inferiority study
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiszasüly mud-pack (Active Comparator): Patients in the Tiszasüly mud-pack group got hot mud-packs for 30 minutes on 10 occasions for 2 weeks (10 working days) on the painful knee.
  Interventions: Other: Tiszasüly hot mud-pack therapy
- Kolop mud-pack (Active Comparator): Patients in the Kolop mud-pack group got hot mud-packs for 30 minutes on 10 occasions for 2 weeks (10 working days) on the painful knee.
  Interventions: Other: Kolop mud-pack

INTERVENTIONS:
Other: Tiszasüly hot mud-pack therapy — Patients received Tiszasüly hot mud-packs (42 Celsius degree) for 30 minutes on 10 occasions for 2 weeks (10 working days) on the painful knee.
  Arms: Tiszasüly mud-pack
Other: Kolop mud-pack — Patients received Kolop hot mud-packs (42 Celsius degree) for 30 minutes on 10 occasions for 2 weeks (10 working days) on the painful knee.
  Arms: Kolop mud-pack

SUMMARY:
In this double-blind, randomized, follow-up study investigators evaluated and compared the effects of Tiszasüly and Kolop mud-pack therapy on pain, function and quality of life in patients with knee osteoarthritis. 30 patients were treated with Tiszasüly hot mud-pack (Group 1), 30 patients with Kolop hot mud-pack (Group 2) for 10 working days. Knee pain, function a nd qualitiy of life were measured at baseline, at the end of treatment and 3 months later.

DETAILED DESCRIPTION:
The aim of this non-inferiority study was to evaluate and compare the effects of Tiszasüly and Kolop mud-pack therapy on pain, function and quality of life in patients with knee osteoarthritis.

Methods: In this double-blind, randomized, follow-up study 60 patients with knee osteoarthritis were treated with either Tiszasüly hot mud-pack (Group 1), or with Kolop hot mud-pack (Group 2) on 10 occasions for 2 weeks (10 working days). 100 mm Visual Analogue Scale (VAS) for knee pain, Western Ontario and McMaster Universities Arthritis Index (WOMAC), Knee Injury and Osteoarthritis Outcome Score (KOOS), Lequesne Index for physical function and EuroQoL-5D for quality-of-life measure were recorded at baseline, at the end of treatment (Week 2) and 3 months later (Week 12).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with knee osteoarthritis (radiologically Kellgren-Laurence II-III. stage)
* resting VAS pain is > 50 mm

Exclusion Criteria:

* infection
* fever
* tumour
* neurologic disorders with numbness and tingling sensation in the lower extremeties
* skin disease aroud the knee
* untreated hypertension
* heart failure (NYHA II-IV. stage)
* inflammatory rheumatic diseases
* knee arthroplasty
* steroid or hialuronic acid injection into the knee joint within 3 months
* physiotherapy of the knee within 3 months
* inflammatory knee osteoarthitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
change in severity of pain at rest | Week 0 and Week 2
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in severity of pain at rest | Week 0 and Week 12
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in function | Week 0 and Week 2
  change from baseline physical function measured by Western Ontario and McMaster Universities Arthritis Index (WOMAC) at week 2. It is comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). All the items are scored on a 100mm visual analogue scale. Values are summed up for a combined WOMAC score. The lower score represents better outcome.
change in function | Week 0 and Week 12
  change from baseline Western Ontario and McMaster Universities Arthritis Index (WOMAC) at week 12. It is comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). All the items are scored on a 100mm visual analogue scale. Values are summed up for a combined WOMAC score. The lower score represents better outcome.
change in function | Week 0 and Week 2
  change from baseline physical function measuredf by Lequesne Index, which is a 10-question survey. It has five questions pertaining to pain or discomfort, 1 question dealing with maximum distance walked, and four questions about activities of daily living.
change in function | Week 0 and Week 12
  change from baseline physical function measured by Lequesne Index, which is a 10-question survey. It has five questions pertaining to pain or discomfort, 1 question dealing with maximum distance walked, and four questions about activities of daily living.
change in function | Week 0 and Week 2
  change from baselilne physical function measured by Knee Injury and Osteoarthritis Outcome Score (KOOS). It is an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in knee osteoarthritis. It has five separately scored subscales: pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec), and knee-related quality of life (QOL). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
change in function | Week 0 and Week 12
  change from baselilne physical function measured by Knee Injury and Osteoarthritis Outcome Score (KOOS). It is an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in knee osteoarthritis. It has five separately scored subscales: pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec), and knee-related quality of life (QOL). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
change in quality of life | Week 0 and Week 2
  change from baseline qualiity of life measured by EuroQoL-5D. It has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), where patients are asked to rate their health problems at five levels (no problems, slight problems, moderate problems, severe problems, extreme problems). It also includes a self-rating of health status on a visual analogue scale (EQ VAS) ranging from 0 to 100 (where 0 means the worst and 100 means the best health status).
change in quality of life | Week 0 and Week 12
  change from baseline qualiity of life measured by EuroQoL-5D. It has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), where patients are asked to rate their health problems at five levels (no problems, slight problems, moderate problems, severe problems, extreme problems). It also includes a self-rating of health status on a visual analogue scale (EQ VAS) ranging from 0 to 100 (where 0 means the worst and 100 means the best health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Petz Aladár County Teaching Hospital, Győr, Hungary